CLINICAL TRIAL: NCT01736774
Title: A Randomized Controlled Trial of Exercise and Manipulative Therapy for Older Persons With Frequent Intermittent Headaches Associated With Neck Pain and Impairment
Brief Title: Exercise and Manipulative Therapy for Older Persons With Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Sureeporn Uthaikhup, Principal Investigator, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRG5580145
Record Dates: First submitted 2012-11-22; First posted 2012-11-29 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Headache
Keywords: Manual therapy; Exercise
MeSH Terms: conditions — Headache; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care intervention (Experimental): Primary care as required including medication
  Interventions: Other: Usual care intervention
- Physiotherapy treatment (Experimental): Exercise and manipulative therapy
  Interventions: Other: Physiotherapy treatment

INTERVENTIONS:
Other: Usual care intervention — The usual care intervention will include appropriate primary care as required including medication
  Arms: Usual care intervention
Other: Physiotherapy treatment — Exercise and manipulative therapy treatment for 10 weeks:The treatment intervention consists of two visits per week for the first four weeks (8 treatments) and one visit per week for the last six weeks (6 treatments)
  Arms: Physiotherapy treatment

SUMMARY:
The presence of cervical musculoskeletal impairment is not specific to cervicogenic headache but other various frequent intermittent headache types (i.e. migraine and tension-type headache) in the elderly population. There has been no trial to date which has investigated the effectiveness of physiotherapy treatment specifically for older persons with various types of headache with associated neck pain and cervical musculoskeletal impairment. Thus, the purpose of study investigate the efficacy of physiotherapy treatment for older persons who have headache concomitant with neck pain and musculoskeletal impairment

DETAILED DESCRIPTION:
Headache is a common health problem that affects quality of life in an older population and imposes substantial economic costs. Headache changes with age. Features of headache become less typical and neck pain is more frequently associated with headache in older persons. We recently demonstrated that the presence of cervical musculoskeletal impairment is not specific to cervicogenic headache (headache caused by the neck). Rather it was present in various frequent intermittent headache types in elders when compared to elders without headache. Changes in headache characteristics with age play an important role not only in diagnosis but also in treatment choice. Impairment in cervical musculoskeletal function found in older persons with headache has implications for headache management choices as the evidence indicates that physiotherapy management methods such as manual therapy and therapeutic exercise are an effective management approach for headache associated with the neck. Physiotherapy treatment would be a safe therapeutic option and may have a beneficial effect for elders with headache who have neck pain and concomitant cervical musculoskeletal dysfunction. This is particularly relevant as there are widespread concerns about medication overuse, adverse drug events and drug interactions in older persons. The effective management of older persons with headache in particular of those with atypical features of headache remains a challenge. Physiotherapy is indicated in those older persons diagnosed with cervicogenic headache but could also be adjunct treatment for those with cervical musculoskeletal signs who are suspected of having transitional headache. At present, there has been no trial to date which has investigated the effectiveness of physiotherapy treatment specifically for older persons with various types of headache with associated neck pain and cervical musculoskeletal impairment. A clinical trial of treatment of cervical musculoskeletal impairment in older persons with various headache types may help guide management of headache in attempts to lesson medication use and cost in this population. Physiotherapy management may be a worthy treatment option particularly in older persons with headache who do not respond well to medication.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers suffering from frequent intermittent headache (either migraine, tension-type headache or cervicogenic headache) at least one per month over a period of 3 months or longer
* Aged 50 years or older, female or male
* A score of ≥ 3/10 on visual analogue scale (VAS) of neck pain
* Evidence of cervical musculoskeletal impairment: restriction in active range of cervical motion in extension and rotation and join tenderness in at least one of the upper joint as detected by manual palpation

Exclusion Criteria:

* Headache diagnosed as following: temporal arteritis, trigeminal neuralgia, cluster headache, chronic paroxysmal hemicrania/hemicranias continua, temporomandibular joint dysfunction
* Other diagnosed disorders: cerebrovascular disease, Parkinson disease, cognitive disturbance
* Previous history of head or neck surgery
* Lack of willingness to receive either pragmatic treatment or usual care
* Physiotherapy or chiropractic treatment for headache in previous 6 months

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Headache frequency | Change from baseline in headache frequency at week 11 and 6 months after intervention
  The number of headache frequency in the past week

SECONDARY OUTCOMES:
Headache intensity | Change from baseline in headache intensity at week 11 and 6 months after intervention
  An average intensity in the past week will be rated on a 1-10 VAS
Headache duration | Change from baseline in headache duration at week 11 and 6 months after intervention
  The number of hours of headache in the past week
Neck pain intensity | Change from baseline in neck pain intensity at week 11 and 6 months after intervention
  Intensity of neck pain will be measured using a 1-10 VAS
Neck pain and disability | Change from baseline in neck pain and disability at week 11 and 6 months after intervention
  Neck pain and disability will be measured using neck disability index (NDI-Thai version)
Quality of life | Change from baseline in quality of life at week 11 and 6 months after intervention
  The Quality of life will be measured using SF-36 (Thai version)
Medication intake | Change from baseline in medication intake at week 11 and 6 months after intervention
  type and dose of all medications taken by subjects will be recorded one week at baseline and prior to follow-up points on a medication diary
Global assessment of treatment benefit | Changes from baseline in global assessment of treatment benefit at week 11 and 6 months after intervention
  Patients perceived benefit of treatment will be measured on a scale from 0 (no benefit) to 10 (maximum benefit)

CONTACTS AND LOCATIONS:
Overall Officials: Sureeporn Uthaikhup, Ph.D., Principal Investigator — Department of Physical Therapy, Faculty of Associated Medical Sciences
Locations (1):
- Department of Physical Therapy, Faculty of Associated Medical Sciences, Chiang Mai, Thailand